CLINICAL TRIAL: NCT05187715
Title: To Study the Safety and Efficacy of Simvastatin in Patients With Hepatopulmonary Syndrome in Cirrhosis- A Double Blind Randomized Controlled Trial
Brief Title: To Study the Safety and Efficacy of Simvastatin in Patients With Hepatopulmonary Syndrome in Cirrhosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-46
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-10

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin with Standard Medical Treatment (Experimental): Simvastatin 40mg OD plus standard treatment plus standard treatment (excluding Pentoxiphylline)
  Interventions: Drug: Simvastatin 40mg; Other: Standard medical Treatment
- Placebo with Standard Medical Treatment (Active Comparator): Matched placebo plus standard treatment (excluding Pentoxiphylline)
  Interventions: Other: Placebo; Other: Standard medical Treatment

INTERVENTIONS:
Drug: Simvastatin 40mg — Simvastatin 40mg OD
  Arms: Simvastatin with Standard Medical Treatment
Other: Placebo — Placebo
  Arms: Placebo with Standard Medical Treatment
Other: Standard medical Treatment — Standard medical Treatment eccluding pentoxiphylline

SUMMARY:
Hepatopulmonary syndrome (HPS) is a frequent pulmonary complication of end-stage liver disease that is characterized by decreased arterial oxygenation caused by intrapulmonary vascular dilatation. Due to the different diagnostic criteria used in different studies, its prevalence ranges from 4% to 47% in patients with cirrhosis. Main underlaying pathogensis for HPS being activation of macrophages which are responsible for iNOS, PDGF and VEGF release contributing to development of intrapulmonary vascular dilatation(IPVD) , and neoangiogenesis leading to anatomical shunt resulting decreased oxygenation. Sphingosine 1 phosphate (S1P) is an essential compound produced and secreted by endothelial cells, platelets and RBC's. S1P prevents adhesion, transmigration and release of inflammatory mediators from macrophages. S1P levels are decreased in cirrhotics. Simvastatin, a HMG CoA inhibitor has many pleotropic effects, Of which one is by agonizing the S1P response and improving oxygenation in HPS patients. Simvastatin at a optimal dose of 40mg/day for 6months. Pre and post simvastatin treatment related oxygenation changes and concurrently its effect on liver fibrosis will be evaluated.

DETAILED DESCRIPTION:
Methodology:

* Study population:All the consecutive patients of cirrhosis admitted to Hepatology department of ILBS will be evaluated for inclusion.
* Study design: Double Blind randomized control trial: Superiority trial. The study will be conductedin Department of Hepatology ILBS.
* Study period: 2 years
* Sample size:

  * Assuming 40% as the response rate to simvastatin and 1% to standard medical treatment with α 5% , power 80% and superiority marging as 10% ,we need to enroll 36 cases 18 in each arm.Further considering 10% drop rate, decided to enroll 40 cases with 20 randomised to 2 groups using block randomisation method taking block score of 4.It is decided to allocate the cases in 2:1 ratio (Simvastatin 2: 1 Placebo) decided to enroll 45 cases so that 30 in simvastatin arm and 15 in standard medical therapy

(Not on pentoxiphylline) arm with block size 15

* Intervention:

  * Patients to be divided into 2 groups
  * Group A-Simvastatin 40mg OD plus standard treatment
  * Group B-Matched placebo plus standard treatment (excluding Pentoxiphylline)
  * Stopping-rule-Development of drug related side effects
  * Disease progression (Increase in baseline MELD by 4 or >25)
* Monitoring and assessment

  * Patients with known cirrhotics will be enrolled as per inclusion criteria and baseline routine testing with complete blood count, liver and kidney function test, ultrasonography of the abdomen, lipid profile, total CPK, measurement of liver and splenic stiffness.Pulmonary blood at the time of HVPG for endothelin-1 and TNF alpha,Nitric oxide levels,S1P expression,KLF-2 levels.
  * Matched placebo not on pentoxiphylline are included.
  * MELD score and Child score, Arterial blood gas analysis, Pulmonary function test,6 minute walk test,Saline contrast 2D ECHO at baseline and at 6months.
  * Clinical evaluation done monthly. Response at the end of 6months.
  * Hepatic venous pressure gradient (HVPG):
  * Prior to the HVPG measurement, a venous access was performed under ultrasonography after local anesthesia. The Seldinger technique was used to insert a catheter into the right brachial vein or the right internal jugular vein. An occlusion balloon catheter of 6 F was guided in a branch of the hepatic veins, usually the median or right vein, under fluoroscopic control and continuous electrocardiographic and pressure monitoring.
  * After inflating the balloon at the catheter's tip (maximum diameter ranges from 8.5-11.5 mm), a venous check was performed to demonstrate complete vessel occlusion. The wedged hepatic vein pressure (WHVP) was measured in this condition. Following that, the free hepatic vein pressure (FHVP) was measured after deflating the balloon at the catheter's tip. On a multi-channel recorder, a permanent trace was obtained. Pressures were also achieved in the inferior vena cava and the right atrium. According to the Baveno VI consensus, the HVPG-response was defined as a 20% or 12 mmHg reduction in HVPG after NSBB treatment.
  * HVPG= WHVP - FHVP (Normal is <5mm of Hg)
  * Ultrasonography of the abdomen:
  * dilated portal vein (>13 mm): non-specific
  * biphasic or reverse flow in portal vein (late stage): pathognomonic
  * recanalization of paraumbilical vein: pathognomonic
  * portal-systemic collateral pathways (collateral vessels/varices)
  * splenomegaly
  * ascites
  * The damping index (showing changes in the doppler hepatic vein waveform) corresponds with hemodynamically significant portal hypertension and HVPG values (together with HVPG changes after treatment)
  * splenic arterial resistive index

Liver and splenic stiffness:

* A 3.5-MHz ultrasound transducer probe is mounted on the axis of a vibrator in the FibroScan device. Mild amplitude, low-frequency (50 Hz) vibrations are transmitted to the liver tissue, causing an elastic shear wave to propagate through the underlying tissue. If the success rate was greater than 60% and the interquartile range (IQR) was greater than 30% of the median value, LS values were accepted.
* Guidelines for measuring SS is same as LS. SS was performed on a supine patient with maximal abduction of the left arm, with the probe positioned in an intercostal space where the spleen was correctly visualized by US. Furthermore, in accordance with the FibroScan's technical features, patients with a splenic parenchymal thickness of >4 cm under the probe were excluded.

  - STATISTICAL ANALYSIS:
* For comparison of parameters pretherapy and posttherapy, the Wilcoxon signed rank test was used. P.05 was considered significant. SPSS version 15.0 statistical software (SPSS Inc, Chicago, Illinois) was used for analysis.

  * Adverse effects:
  * 1. Major Sideeffects of Simvastatin
  * Rhabdomyolysis(Raised Total CPK > 3ULN)
  * Bradycardia
  * Transaminitis (ALT >5ULN)
  * Headache
  * Constipation
  * Upper respiratory tract infection

    2. HVPG related complications
  * Transient arrhythmias
  * Vagal reaction
  * Local access pain and bleeding
  * Stopping rule :
* Development of serious adverse effects leading to withdrawal of the drug or death from any cause.
* Disease progression (Increase in baseline MELD by 4 or >25)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed case of Hepato-pulmonary syndrome AaPO2 > 15 mm Hg on standing room air arterial blood gas (ABG). PaO2<80 mmHg for clinical HPS between 18-70 years of years
2. Child A/B cirrhosis, Child C with CTP score of =/<10
3. Patient with no liver transplant option

Exclusion Criteria:

1. Child-C cirrhosis CTP >10
2. Very Severe HPS
3. Acute-on-chronic liver failure
4. Thrombosis of splenoportal axis
5. Hepatocellular carcinoma
6. Renal dysfunction
7. Patients intolerant to beta blockers (history of hypotension or bradycardia)
8. Contraindication for beta-blockers (history of chronic obstructive pulmonary disease, atrioventricular block)
9. Pregnant females
10. Refusal to participate in the study
11. Hepatic Hydrothorax

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-02-26 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Achievement of complete response by the end of 6 months | 6 months

SECONDARY OUTCOMES:
Transplant free survival | 3 months
Transplant free survival | 6 months
Severity of Liver Disease | 6 months
  Severity will be assess by MELD Na (Model for End Stage Liver Disease)
Development of serious adverse effects leading to withdrawal of the drug or death from any cause. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided